CLINICAL TRIAL: NCT05142215
Title: ORBITA-CTO Pilot: A Comparison of the Impact of CTO PCI Versus Placebo on Angina in Patients With Background Optimal Medical Therapy - a Pilot Study
Brief Title: A Placebo-controlled Trial of Chronic Total Occlusion Percutaneous Coronary Intervention for the Relief of Stable Angina
Acronym: ORBITA-CTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299940
Record Dates: First submitted 2021-11-09; First posted 2021-12-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stable Angina; Chronic Total Occlusion of Coronary Artery
Keywords: Angina; Chronic total occlusion; Angioplasty
MeSH Terms: conditions — Angina, Stable; Angina Pectoris | interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percutaneous coronary intervention (Active Comparator): Percutaneous coronary intervention (PCI) for chronic total occlusion (CTO).
  Interventions: Procedure: Percutaneous coronary intervention
- Placebo percutaneous coronary intervention (Placebo Comparator): Placebo procedure for chronic total occlusion (CTO).
  Interventions: Procedure: Placebo percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention using drug eluting stents and contemporary CTO PCI techniques on background of optimal medical therapy.
  Other Names: Coronary angioplasty
  Arms: Percutaneous coronary intervention
Procedure: Placebo percutaneous coronary intervention — Placebo percutaneous coronary intervention procedure on background of optimal medical therapy.
  Arms: Placebo percutaneous coronary intervention

SUMMARY:
ORBITA-CTO Pilot is a double blinded randomised placebo-controlled trial comparing the effects of chronic total occlusion percutaneous coronary intervention versus placebo on symptoms of angina in patients with background optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

ORBITA CTO will enrol patients who meet all 5 of the following criteria:

1. Accepted for CTO PCI procedure by a specialist CTO operator.
2. Patients with symptoms related to a single vessel CTO (≥3 months duration, or probable CTO where duration is unknown) in a vessel of at least 2.5mm diameter without angiographically significant (LMS ≥50%, LAD/Cx/RCA/Graft ≥70%, ≥2mm diameter) coronary artery stenosis in remaining non-CTO vessels.

   Symptoms are:

   a) Typical exertional angina defined as: i) constricting discomfort in the front of the chest or in the neck, jaw, shoulder or arm ii) precipitated by physical exertion iii) relieved by rest or nitrates within 5 minutes b) Angina symptoms at rest (including decubitus angina and post-prandial angina).

   c) Shortness of breath on exertion considered to be angina equivalent.
3. Clinical evidence of ischaemia in CTO territory on dobutamine stress echocardiography, nuclear myocardial perfusion scan, stress perfusion CMR or PET).
4. Evidence of viability: If left ventricular angiogram or echocardiogram demonstrates LV impairment or RWMA then viability must be demonstrated.
5. J-CTO score ≤ 3.

Exclusion Criteria:

1. Acute coronary syndrome within 4 weeks.
2. PCI to non-CTO lesion in prior 4 weeks as part of ACS or elective PCI.
3. Non-revascularised clinically important non-CTO vessel.
4. Proven ischaemia (invasive or non-invasive) in non-culprit territory.
5. Contraindications to PCI or drug-eluting stent (DES) implantation.
6. Inability to tolerate or contraindication to DAPT.
7. Severe valvular heart disease.
8. Severe chronic pulmonary disease (FEV1 <30% of predicted value).
9. Severe musculoskeletal disease resulting in immobility.
10. Life expectancy <2years.
11. Pregnancy.
12. Age <18years.
13. Inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change in angina symptom ordinal scale score between groups | 24 & 26 weeks
  Change in angina symptom ordinal scale score between groups

SECONDARY OUTCOMES:
Physical limitation, angina frequency, angina stability, treatment satisfaction and quality of life scores as measured by the Seattle Angina Questionnaire (SAQ) | 24 & 26 weeks
  Physical limitation, angina frequency, angina stability, treatment satisfaction and quality of life scores as measured by the Seattle Angina Questionnaire (SAQ)
SAQ summary score | 24 & 26 weeks
  SAQ summary score
Quality of life as measured by EQ-5D-5L | 24 & 26 weeks
  Quality of life as measured by EQ-5D-5L
Change in Rose dyspnea scale | 24 & 26 weeks
  Change in Rose dyspnea scale
Change in peak VO2 and VO2 at AT | 24 weeks
  Change in peak VO2 and VO2 at AT
Fidelity of blinding using Bang's blinding index (BI) | 24 weeks
  Fidelity of blinding using Bang's blinding index (BI)
Protocol adherence | 26 weeks
  Proportion of participants adherent to allocated randomised treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Davies, MRCP PhD, Principal Investigator — Essex Cardiothoracic Centre, UK; Sarosh Khan, MRCP, Study Director — Essex Cardiothoracic Centre, UK
Locations (3):
- United Kingdom (3):
  - Essex Cardiothoracic Centre, Basildon, Essex
  - Royal Bournemouth Hospital, Bournemouth
  - St. George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No